CLINICAL TRIAL: NCT03914092
Title: Intralesional Steroid Injection Versus Accent Method of Voice Therapy in Management of Vocal Nodules: A Randomized Controlled Trial
Brief Title: Intralesional Steroid Injection Versus Voice Therapy in Management of Vocal Nodules
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Nada Ali Kamel, principle investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: QWE
Record Dates: First submitted 2019-04-06; First posted 2019-04-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2025-07

CONDITIONS: Vocal Nodules in Adults
MeSH Terms: interventions — Triamcinolone Acetonide

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group (Experimental): female patients with vocal fold nodules undergoing intralesional steroid injection
  Interventions: Drug: triamcinolone acetonide injection
- control group (Active Comparator): female patients with vocal fold nodules undergoing Smith Accent voice therapy
  Interventions: Behavioral: Smith Accent method of voice therapy

INTERVENTIONS:
Drug: triamcinolone acetonide injection — 0.1- 0.3 mm percutaneous intralesional injection
  Other Names: Epirelefan
  Arms: study group
Behavioral: Smith Accent method of voice therapy — regular sessions of smith accent voice therapy (about 24 sessions, twice session / week) for 3 months
  Arms: control group

SUMMARY:
Vocal nodules represent 16 % of benign vocal fold lesions.They are caused by chronic voice abuse or misuse and often occur in children and adult females. The resultant dysphonia leads to personal, social and occupational problems.

The first line of treatment is voice rest and voice therapy. The Accent method is a holistic technique for behavior readjustment voice therapy which targets various voice parameters as loudness, pitch and timbre. However, voice rest and voice therapy are sometimes difficult to be carried out in patients with voice-related occupations. So, complete resolution may not be possible in all patients. When voice therapy is inefficient, resection is performed by laryngeal microsurgery under general anesthesia. However, the role of surgery is much restricted.

DETAILED DESCRIPTION:
An intralesional steroid injection to vocal nodules has come to the forefront as another treatment choice. Steroids decrease the synthesis and maturation of collagen, suppress fibroblast function, and inhibit the antibacterial phagocytic action of some defense cells and vasoactive substances release.These actions are considered to be functional for treating vocal nodules. Many studies, investigated steroid injection in benign lesions including nodules, reported that 93-100% of the nodules either disappeared or improved. The reported nodules recurrence rate after 2 years was 26.7- 31%.

However, to our knowledge, no previous study has compared vocal nodule steroid injection with a group receiving voice therapy to accurately assess the clinical role of vocal fold steroid injection.

ELIGIBILITY:
Inclusion Criteria:

- 1- Female patients diagnosed with bilateral vocal fold soft edematous nodules with preserved or minimally impacted stroboscopic waves , don't exceed base 2.5 mm and apex .5mm.

2- age: 18-55 years. 3- Normal articulation, resonance and language ability. 4- Normal hearing.

Exclusion Criteria:

* 1- Previous voice therapy or micro-phono-surgery. 2- Use of drugs (which may cause changes in laryngeal function, mucosa, or muscle activity).

  3- History of allergies, lung disease, gastroesophageal reflux disease, or other concomitant vocal pathology (e.g., vocal polyp and vocal cyst).

  4- Current psychiatric, neurological conditions.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2019-06-29 (Actual); Primary Completion 2022-08-15 (Actual); Study Completion 2023-08-28 (Actual)

PRIMARY OUTCOMES:
Subjective measurements of severity of dysphonia | Before intervention
  Measurements of change of Grade of Dysphonia, Roughness, Breathiness, Asthenia, and Straining by auditory perceptual assessment using the GRBAS scale. Grades ranging from 0 (normal) up to 3 (severe)
Subjective measurements of patient's assessment of voice severity | Before intervention
  Measurements of scores of Arabic Voice Handicap Index
Objective measurements of vocal nodules size | before intervention
  Measurements of base and rise of nodules using videostroboscopic examination
Objective measurements of vocal pitch | Before intervention
  Measurements of acoustic analysis: fundamental frequency (Hz)
Objective measurements of vocal waveform frequency aperiodicity | Before intervention
  Measurements of acoustic analysis: jitter (%)
Objective measurements of vocal waveform amplitude aperiodicity | Before intervention
  Measurements of acoustic analysis: shimmer (dB)
Objective measurements of vocal waveform periodicity to aperiodicity ratio | Before intervention
  Measurements of acoustic analysis : harmonic to noise ratio(dB)
Objective measurements of glottal efficiency | Before intervention
  Measurements of aerodynamic parameter : Maximum phonation time (seconds)

SECONDARY OUTCOMES:
Change in Subjective measurements of severity dysphonia | 1 week and 1, 2, 3, and 6 months after intervention
  Measurements of change of Grade of Dysphonia, Roughness, Breathiness, Asthenia, and Straining by auditory perceptual assessment using the GRBAS scale. Grades ranging from 0 (normal) up to 3 (severe)
Change in subjective measurements of patient's assessment of voice severity | 1 week and 1, 2, 3 and 6 months after intervention
  Measurements of change in scores of Arabic Voice Handicap Index
Change in objective measurements of vocal nodules size | 1 week and 1, 2, 3 and 6 months after intervention
  Measurements of change in base and rise of nodules using videostroboscopic examination
Change in objective measurements of vocal pitch | 1 week and 1, 2, 3 and 6 months after intervention
  Measurements of change in acoustic analysis including fundamental frequency (Hz)
Change in objective measurements of vocal waveform frequency aperiodicity | 1 week and 1, 2, 3 and 6 months after intervention
  Measurements of change in acoustic analysis : jitter (%)
Change in objective measurements of vocal waveform amplitude aperiodicity | 1 week and 1, 2, 3 and 6 months after intervention
  Measurements of change in acoustic analysis : shimmer (dB)
Change in objective measurements of vocal waveform periodicity to aperiodicity ratio | 1 week and 1, 2, 3 and 6 months after intervention
  Change in measurements of acoustic analysis : harmonic to noise ratio (dB)
Change in objective measurements of glottal efficiency | 1 week and 1, 2, 3 and 6 months after intervention
  Measurements of change in aerodynamic parameter: Maximum phonation time (seconds)

CONTACTS AND LOCATIONS:
Overall Officials: Nada A Kamel, M.Sc., Principal Investigator — Assiut University
Locations (1):
- Assiut university hospitals, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bassiouny S. Efficacy of the accent method of voice therapy. Folia Phoniatr Logop. 1998;50(3):146-64. doi: 10.1159/000021458. PMID 9691529
- [Background] Tateya I. Laryngeal steroid injection. Curr Opin Otolaryngol Head Neck Surg. 2009 Dec;17(6):424-6. doi: 10.1097/MOO.0b013e3283327d4c. PMID 19779349
- [Background] Campagnolo AM, Tsuji DH, Sennes LU, Imamura R, Saldiva PH. Histologic study of acute vocal fold wound healing after corticosteroid injection in a rabbit model. Ann Otol Rhinol Laryngol. 2010 Feb;119(2):133-9. doi: 10.1177/000348941011900211. PMID 20336925
- [Background] Lee SH, Yeo JO, Choi JI, Jin HJ, Kim JP, Woo SH, Jin SM. Local steroid injection via the cricothyroid membrane in patients with a vocal nodule. Arch Otolaryngol Head Neck Surg. 2011 Oct;137(10):1011-6. doi: 10.1001/archoto.2011.168. PMID 22006779
- [Background] Woo JH, Kim DY, Kim JW, Oh EA, Lee SW. Efficacy of percutaneous vocal fold injections for benign laryngeal lesions: Prospective multicenter study. Acta Otolaryngol. 2011 Dec;131(12):1326-32. doi: 10.3109/00016489.2011.620620. PMID 22074107
- [Background] Wang CT, Lai MS, Hsiao TY. Comprehensive Outcome Researches of Intralesional Steroid Injection on Benign Vocal Fold Lesions. J Voice. 2015 Sep;29(5):578-87. doi: 10.1016/j.jvoice.2014.11.002. Epub 2015 May 2. PMID 25944294
- [Background] Wang CT, Lai MS, Cheng PW. Long-term Surveillance Following Intralesional Steroid Injection for Benign Vocal Fold Lesions. JAMA Otolaryngol Head Neck Surg. 2017 Jun 1;143(6):589-594. doi: 10.1001/jamaoto.2016.4418. PMID 28334309